CLINICAL TRIAL: NCT06575634
Title: Effects of Supervised Exercise on Rheological Functions of Erythrocyte in Patients With End-Stage Renal Disease on Hemodialysis
Brief Title: Exercise Therapy on Rheological Functions of Erythrocyte in Hemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102279A3101
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis Complication
Keywords: Hemodialysis; Exercise training; Erythrocyte; Rheology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise training (Experimental)
  Interventions: Behavioral: Supervised exercise training
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Supervised exercise training — Participants perform Intradialytic cycling exercise training in the hospital for 6 months (24 weeks) and 3 months (12 weeks) at home. Exercise prescription: 50-60% maximal workload for 20-30 minutes, including low intensity warm-up and cool down (30% of maximal workload).
  Arms: Supervised exercise training

SUMMARY:
To improve aerobic capacity, muscular function, and health-related quality of life in patients with end-stage renal disease (ESRD), regular exercise is recommended. Supervised intradialytic exercise at moderate intensity is a viable approach to ensure patient safety, maintain compliance, and effectively enhance physiological adaptations. However, the impact of exercise training on erythrocyte rheological properties in ESRD patients, such as red blood cell deformability, aggregation, and oxygen transport capacity, remains unclear.

Method: ESRD patients (anticipated n=180) will undergo supervised exercise training therapy three times per week for six months in the hospital, followed by three months at home. Cardiopulmonary exercise tests will be conducted before and after the intervention. Erythrocyte deformability and aggregation will be assessed using a laser-assisted optical rotational cell analyzer (LORCA), while additional protein levels and reactive oxygen species (ROS) status will be measured using a flow cytometer. This will help determine how exercise affects the rheological properties of red blood cells in this population.

DETAILED DESCRIPTION:
Renal dysfunction often stems from cardiovascular-related comorbidities or metabolic disorders, leading to the accumulation of excessive inflammatory products or damaging the bioenergetic health of red blood cells. This eventually contributes to the development of chronic kidney disease (CKD). At the most advanced stage, known as end-stage renal disease (ESRD), patients suffer from severe uremia and renal failure, necessitating renal replacement therapy, typically in the form of dialysis.

Hemodialysis (HD) is the most common treatment for ESRD patients, especially in Taiwan, which has the highest global prevalence of HD due to related chronic diseases and a comprehensive National Health Insurance program. However, long-term maintenance HD is associated with physical inactivity and a low quality of life. As a result, exercise training is recommended to improve physiological adaptations and enhance functional capacity in HD patients. Supervised intradialytic exercise in clinical settings offers a safer and more progressive approach, leading to low dropout rates and better compliance.

Red blood cell dysfunction is a significant issue in ESRD, as impaired red blood cells can affect their deformability, aggregation, and oxygen transport capacity.

The purpose of this study is to establish reliable measurements of red blood cell function in HD patients and assess cardiovascular and muscular fitness, along with the effects of intradialytic exercise on these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis and medication at least for 6 weeks
* Kt/V score > 1.2

Exclusion Criteria:

* Under 20 years-old
* Hyperkalemia occurs within 3 month
* Having orthopedic or muscular diseases
* Other concerned medical, psychological or physiological diseases
* Pregnancy
* Other exercise contraindications

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Deformability of erythrocytes | 9 months
  Red blood cells (RBCs) deformability refers to the cells' ability to adapt their shape to the dynamically changing flow conditions so as to minimize their resistance to flow.
Aggregation of erythrocytes | 9 months
  Erythrocyte aggregation is the reversible clumping of red blood cells (RBCs) under low shear forces or at stasis.

SECONDARY OUTCOMES:
Cardiopulmonary fitness | 9 months
  ESRD patients performed cardiopulmonary exercise testing (CPET) to assess their aerobic capacity. CPET composed of continuous workload increment of 10 W/min until exhaustion (usually within 8-12 minutes). Oxygen consumption, carbon dioxide production, ventilation, respiratory rate would be recorded.
Quality of life in ESRD patients | 9 months
  The investigators would use a qusionnaire, The Kidney Disease Quality of Life 36-item short form survey (KDQOL-36), to record and scale the qulaity of life in ESRD patients. The KDQOL-36 (Kidney Disease Quality of Life 36-Item Short Form Survey) measures the quality of life in kidney disease patients. It uses a score range from 0 to 100, where higher scores indicate better quality of life and lower scores indicate worse outcomes. Ensure to note this when reporting results to clarify that higher scores reflect fewer symptoms and better overall well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Shyan Wang, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No